CLINICAL TRIAL: NCT06511167
Title: National, Prospective, Multicentre Post Market Surveillance Study on "Patient Reported Outcome" of Implant Based Primary or Secondary Reconstructive Breast Surgery After Mastectomy Using the Complete Resorbable Synthetic TIGR® Matrix
Brief Title: Post-market Surveillance Study to Evaluate the Quality of Life and the Safety and Effectiveness of the TIGR® Matrix After Reconstructive Breast Surgery
Acronym: TIGR-Matrix
Status: Recruiting | Type: Observational
Sponsor: AWOgyn (Other)
Collaborators: Esculape GmbH (Unknown)
Responsible Party: Sponsor
Other Study IDs: AWO-001
Record Dates: First submitted 2024-07-16; First posted 2024-07-19 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Implant Based Breast Reconstruction
Keywords: TIGR® Matrix; Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: TIGR® Matrix — bioresorbable, synthetic, surgical mesh

SUMMARY:
The goal of this observational study is to evaluate the quality of life of participants who have undergone implant-based breast surgery. This will be done using the BREAST-Q questionnaire. The study also aims to demonstrate that the fully resorbable TIGR® Matrix is safe and effective.

DETAILED DESCRIPTION:
This national, multicentre, prospective, non-randomized post market surveillance clinical device investigation will be performed to obtain information on the resorbable surgical mesh TIGR® Matrix used during an implant-based breast surgery. Data will be collected on the participants' quality of life as well as on the rate of complications of the device under investigation.

ELIGIBILITY:
Inclusion Criteria:

* Women with histologically confirmed breast cancer or precancerosis or genetic pre- existing conditions with increased risk of breast cancer or with a family history all with an indication for skin sparing or nipple sparing mastectomy (SSM or NSM); or women with indication of prophylactic operation
* The health of women must comply with ECOG performance status 0-2
* The decision for the implementation of the TIGR® Matrix was made before and independently from study enrollment
* Participant is mentally able to understand the nature, aims, or possible consequences of the clinical investigation
* Patient information has been handed out and subject signed informed consent
* Participant has attained full age of 18 years

Exclusion Criteria:

* Pregnancy or breast-feeding patients
* Known intolerance to the material, mesh-implants under investigation
* Metastatic breast cancer (with a life expectancy < 5 years)
* Medicinal dis-regulated diabetes
* Inadequate bone marrow function with neutrophil granulocytes<1500 and blood plates < 100.000/µl
* Lack or withdrawn of written patients informed consent
* Lack of patient compliance regarding data collection, treatment or follow-up investigations in the scope of the protocol
* Participant is institutionalized by court or official order (MPDG §27)
* Participation in another surgical clinical investigation that influence the surgical technique or outcome.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women who will undergo breast prepectoral implant-based breast reconstructive surgery
Sampling Method: Non-Probability Sample
Enrollment: 135 (Estimated)
Dates: Start 2024-11-08 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Quality of Life 12 months after surgery (BREAST-Q) | 12 months after surgery
  Quality of Life will be assessed using the validated Breast-Q patient-reported outcome measure in order to compare the presence, severity and impact of the participants' symptoms on their quality of life and daily activities

SECONDARY OUTCOMES:
Quality of Life 6, 24, 36 months after surgery (BREAST-Q) | 6, 24, 36 months after surgery
  Quality of Life will be assessed using the validated Breast-Q patient-reported outcome measure in order to compare the presence, severity and impact of the participants' symptoms on their quality of life and daily activities
Complication rate | minimum of 3 years and a maximum of 5 years after surgery
  The number and rate of occurrence of major complications, minor complications; Serious Adverse Events (SAEs) and Adverse Events (AEs)
Complication rate of specific complications | minimum of 3 years and a maximum of 5 years after surgery
  Complication rate of:
  * Seroma-Volume (Sum of fluid-volume during the drainage-time)
  * Need for aspiration in symptomatic patients, number of aspirations in postoperative follow up
  * Reconstructive failure (defined as unplanned implant loss)
Days with drain(s) | during hospital stay after surgery
  The number of days between placement of drain system and removal of the drain
Days of hospital stay | surgery to discharge from hospital
  The number of days the participant spend in hospital after surgery
Cosmetic outcome | 6, 12, 24 ,36 month after surgery
  Domains of cosmesis of BREAST-Q as perceived by the participant as well as perceived by the physician
Rate of unplanned conversion operations | minimum of 3 years and a maximum of 5 years after surgery
  Rate of unplanned conversion operations (to mastectomy without reconstruction; to mastectomy with reconstruction; to autologous reconstruction)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Thill, Prof., Study Chair — AWOgyn
Locations (5):
- Germany (5):
  - GRN-Klinik Weinheim, Weinheim, Baden-Wurttemberg
  - Klinik und Poliklinik für Frauenheilkunde Technische Universität München, München, Bavaria
  - Agaplesion Markus Krankenhaus Frankfurt, Frankfurt am Main, Hesse
  - Evangelisches Krankenhaus Wesel, Wesel, North Rhine-Westphalia
  - Krankenhaus St. Elisabeth und St. Barbara Halle (Saale) GmbH, Halle